CLINICAL TRIAL: NCT00003424
Title: Randomised Trial of Tamoxifen Versus Placebo for the Treatment of Inoperable Hepatocellular Carcinoma
Brief Title: Tamoxifen in Treating Patients With Primary Liver Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Medical Research Council (NMRC), Singapore (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NMRC-AHCC01; CDR0000066444 (Registry Identifier: PDQ (Physician Data Query)); EU-98018
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-08

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Tamoxifen

INTERVENTIONS:
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of cancer cells. Hormone therapy using tamoxifen may fight liver cancer by blocking the absorption of estrogen. It is not yet known whether receiving tamoxifen is more effective than no further therapy in treating patients with primary liver cancer.

PURPOSE: Randomized phase III trial to compare high-dose tamoxifen with no further treatment in treating patients with liver cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic role of tamoxifen in patients with inoperable hepatocellular carcinoma in terms of overall survival and quality of life.

OUTLINE: This is a randomized, double blind, placebo controlled study of tamoxifen. Patients are randomized to one of 3 treatment arms. Arm I: Patients receive placebo orally twice daily for one year. Arms II and III: Patients receive tamoxifen, at 1 of 2 different doses, orally twice daily for one year. Quality of life is assessed before treatment and then monthly thereafter. Patients are followed monthly until death.

PROJECTED ACCRUAL: This study will accrue 300 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or radiologically confirmed inoperable hepatocellular carcinoma Serum alfa-feto protein level at least 500 ug/L OR Positive lipiodol uptake

PATIENT CHARACTERISTICS: Age: 10 to 90 Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine less than 1.7 mg/dL Other: No encephalopathy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemoembolization therapy for disease No prior systemic chemotherapy for disease Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: No prior surgery for disease Other: No prior percutaneous injection

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1997-04; Primary Completion 2000-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, MBBS, FRCS, FAMS, Study Chair — National Cancer Centre, Singapore
Locations (8):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- University of Udayana, Sanglah, Denpasar, Bali, Indonesia
- Universiti Kebangsaan Malaysia, Bangi, Malaysia
- Wellington Cancer Centre, Wellington, New Zealand
- Pakistan (2):
  - National Cancer Institute - Karachi, Karachi
  - Nishtar Medical College, Multan, Multan
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - National Cancer Centre - Singapore, Singapore